CLINICAL TRIAL: NCT01779375
Title: Restoring Insulin Secretion Pediatric Medication Study
Brief Title: RISE Pediatric Medication Study
Acronym: RISE Peds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RISE Study Group (Network)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RISE Pediatric; 5U01DK094406-02 (NIH)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Prediabetes; Type 2 Diabetes
Keywords: Children; Pediatric
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin alone (Active Comparator): Metformin will be titrated to the maximum dose tolerated (up to 2000 mg/day).
  Interventions: Drug: Metformin
- Glargine followed by Metformin (Active Comparator): Basal insulin glargine for 3 months titrated to achieve a morning fasting blood glucose of 85-95 mg/dl, followed by metformin (titrated up to 2000 mg/day) for 9 months.
  Interventions: Drug: Metformin; Drug: Glargine

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage
Drug: Glargine
  Other Names: Insulin glargine, Lantus
  Arms: Glargine followed by Metformin

SUMMARY:
The RISE Pediatric Medication Study is a 2-arm, 4-center, clinical trial of children with prediabetes and early type 2 diabetes to address the hypothesis that aggressive glucose lowering will lead to recovery of beta-cell function that will be sustained after withdrawal of treatment. Pediatric participants (ages 10-19) will be randomized to one of the following treatment regimens: (1) metformin alone or (2) early intensive treatment with basal insulin glargine followed by metformin.

The primary clinical question RISE will address is: Are improvements in ß-cell function following 12 months of active treatment maintained for 3 months following the withdrawal of therapy? Secondary outcomes will assess durability of glucose tolerance following withdrawal of therapy, and whether biomarkers obtained in the fasting state predict parameters of ß-cell function, insulin sensitivity and glucose tolerance and the response to an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting plasma glucose ≥90 mg/dl plus 2-hour glucose ≥140 mg/dl on 75 gm OGTT plus laboratory-based HbA1c ≤8.0% if treatment naïve. There is no upper limit for the 2-hour glucose on OGTT. In those taking metformin laboratory-based HbA1c must be ≤7.5% if on metformin for <3 months and ≤7.0% if on metformin for 3-6 months.
2. Age 10-19 years
3. Pubertal development Tanner stage >1 as defined by breast stage >1 in girls, and testes >3 cc's in boys.
4. Body mass index (BMI) ≥85th percentile but ≤50 kg/m2
5. Self-reported diabetes <6 months in duration
6. Treatment with metformin for <6 months preceding screening

Exclusion Criteria:

1. Underlying disease likely to limit life span and/or increase risk of intervention or an underlying condition that is likely to limit ability to participate in outcomes assessment
2. An underlying disease that affects glucose metabolism other than type 2 diabetes mellitus
3. Taking medications that affect glucose metabolism, or has an underlying condition that is likely to require such medications
4. Treatment with insulin for >1 week preceding screening
5. Active infections
6. Renal disease (serum creatinine >1.2 mg/dl) or serum potassium abnormality (<3.4 or >5.5 mmol/l)
7. Anemia (hemoglobin <11 g/dl in girls, <12 g/dl in boys) or known coagulopathy
8. Cardiovascular disease, including uncontrolled hypertension defined as average systolic or diastolic blood pressure > 99 percentile for age or >135/90, despite adequately prescribed antihypertensive medications. Participants must be able to safely tolerate administration of intravenous fluids required during clamp studies.
9. History of conditions that may be precipitated or exacerbated by a study drug:

   1. Serum alanine transaminase (ALT) more than 3 times the upper limit of normal
   2. Excessive alcohol intake
   3. Sub-optimally treated thyroid disease
10. Conditions or behaviors likely to affect the conduct of the RISE Study

    1. Participant and/or parents unable or unwilling to give informed consent
    2. Participant and/or parents unable to adequately communicate with clinic staff
    3. Another household member is a participant or staff member in RISE
    4. Current, recent or anticipated participation in another intervention research project that would interfere with any of the interventions/outcomes in RISE
    5. Weight loss of ≥5% of body weight in the past 3 months for any reason other than post-partum weight loss. Participants taking weight loss drugs or using preparations taken for intended weight loss are excluded.
    6. Likely to move away from participating clinics in next 2 years
    7. Current (or anticipated) pregnancy and lactation.
    8. A pregnancy that was completed less than 6 months prior to screening.
    9. Breast feeding within 6 months prior to screening.
    10. Women of childbearing potential who are unwilling to use adequate contraception
    11. Major psychiatric disorder that, in the opinion of clinic staff, would impede the conduct of RISE
11. Additional conditions may serve as criteria for exclusion at the discretion of the local site.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2013-06-16 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Childrens Hospital Colorado, Denver, Colorado
  - Yale School of Medicine Pediatric Obesity and Type 2 Diabetes Clinic, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Will share all research data via the NIDDK repository 2 years after final patient visit from the RISE consortium in ~2020. Data may be obtained from the repository directly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Through the NIDDK repository in 2020, indefinitely.
Access Criteria: Following NIDDK repository instructions.

REFERENCES:
- [Background] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: II. Observations Using the Oral Glucose Tolerance Test. Diabetes Care. 2018 Aug;41(8):1707-1716. doi: 10.2337/dc18-0243. Epub 2018 Jun 25. PMID 29941498
- [Background] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: I. Observations Using the Hyperglycemic Clamp. Diabetes Care. 2018 Aug;41(8):1696-1706. doi: 10.2337/dc18-0244. Epub 2018 Jun 25. PMID 29941497
- [Background] Hannon TS, Kahn SE, Utzschneider KM, Buchanan TA, Nadeau KJ, Zeitler PS, Ehrmann DA, Arslanian SA, Caprio S, Edelstein SL, Savage PJ, Mather KJ; RISE Consortium. Review of methods for measuring beta-cell function: Design considerations from the Restoring Insulin Secretion (RISE) Consortium. Diabetes Obes Metab. 2018 Jan;20(1):14-24. doi: 10.1111/dom.13005. Epub 2017 Jun 22. PMID 28493515
- [Background] RISE Consortium. Restoring Insulin Secretion (RISE): design of studies of beta-cell preservation in prediabetes and early type 2 diabetes across the life span. Diabetes Care. 2014;37(3):780-8. doi: 10.2337/dc13-1879. Epub 2013 Nov 5. PMID 24194506
- [Result] RISE Consortium. Impact of Insulin and Metformin Versus Metformin Alone on beta-Cell Function in Youth With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes. Diabetes Care. 2018 Aug;41(8):1717-1725. doi: 10.2337/dc18-0787. Epub 2018 Jun 25. PMID 29941500
- [Derived] Tjaden AH, Edelstein SL, Arslanian S, Barengolts E, Caprio S, Cree-Green M, Lteif A, Mather KJ, Savoye M, Xiang AH, Kahn SE. Reproducibility of Glycemic Measures Among Dysglycemic Youth and Adults in the RISE Study. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1125-e1133. doi: 10.1210/clinem/dgad135. PMID 36938582
- [Derived] Utzschneider KM, Tripputi MT, Kozedub A, Barengolts E, Caprio S, Cree-Green M, Edelstein SL, El Ghormli L, Hannon TS, Mather KJ, Palmer J, Nadeau KJ; RISE Consortium. Differential loss of beta-cell function in youth vs. adults following treatment withdrawal in the Restoring Insulin Secretion (RISE) study. Diabetes Res Clin Pract. 2021 Aug;178:108948. doi: 10.1016/j.diabres.2021.108948. Epub 2021 Jul 15. PMID 34274407
- [Derived] Kahn SE, Edelstein SL, Arslanian SA, Barengolts E, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Mather KJ, Nadeau KJ, Utzschneider KM, Xiang AH, Buchanan TA; RISE Consortium; Rise Consortium Investigators:. Effect of Medical and Surgical Interventions on alpha-Cell Function in Dysglycemic Youth and Adults in the RISE Study. Diabetes Care. 2021 Sep;44(9):1948-1960. doi: 10.2337/dc21-0461. Epub 2021 Jun 16. PMID 34135015
- [Derived] Sam S, Edelstein SL, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Ehrmann DA, Hannon TS, Tjaden AH, Kahn SE, Mather KJ, Tripputi M, Utzschneider KM, Xiang AH, Nadeau KJ; RISE Consortium; RISE Consortium Investigators. Baseline Predictors of Glycemic Worsening in Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes in the Restoring Insulin Secretion (RISE) Study. Diabetes Care. 2021 Sep;44(9):1938-1947. doi: 10.2337/dc21-0027. Epub 2021 Jun 15. PMID 34131048
- [Derived] Kahn SE, Mather KJ, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Nadeau KJ, Utzschneider KM, Xiang AH, Edelstein SL; RISE Consortium; Rise Consortium Investigators:. Hyperglucagonemia Does Not Explain the beta-Cell Hyperresponsiveness and Insulin Resistance in Dysglycemic Youth Compared With Adults: Lessons From the RISE Study. Diabetes Care. 2021 Sep;44(9):1961-1969. doi: 10.2337/dc21-0460. Epub 2021 Jun 15. PMID 34131047
- [Derived] Arslanian SA, El Ghormli L, Kim JY, Tjaden AH, Barengolts E, Caprio S, Hannon TS, Mather KJ, Nadeau KJ, Utzschneider KM, Kahn SE; RISE Consortium. OGTT Glucose Response Curves, Insulin Sensitivity, and beta-Cell Function in RISE: Comparison Between Youth and Adults at Randomization and in Response to Interventions to Preserve beta-Cell Function. Diabetes Care. 2021 Mar;44(3):817-825. doi: 10.2337/dc20-2134. Epub 2021 Jan 12. PMID 33436401
- [Derived] Hannon TS, Edelstein SL, Arslanian SA, Caprio S, Zeitler PS, Buchanan TA, Ehrmann DA, Mather KJ, Tripputi M, Kahn SE, Nadeau KJ; RISE Consortium. Withdrawal of medications leads to worsening of OGTT parameters in youth with impaired glucose tolerance or recently-diagnosed type 2 diabetes. Pediatr Diabetes. 2020 Dec;21(8):1437-1446. doi: 10.1111/pedi.13129. Epub 2020 Oct 13. PMID 32985775
- [Derived] RISE Consortium. Obesity and insulin sensitivity effects on cardiovascular risk factors: Comparisons of obese dysglycemic youth and adults. Pediatr Diabetes. 2019 Nov;20(7):849-860. doi: 10.1111/pedi.12883. Epub 2019 Jul 29. PMID 31301210
- [Derived] RISE Consortium; RISE Consortium Investigators. Effects of Treatment of Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes With Metformin Alone or in Combination With Insulin Glargine on beta-Cell Function: Comparison of Responses In Youth And Adults. Diabetes. 2019 Aug;68(8):1670-1680. doi: 10.2337/db19-0299. Epub 2019 Jun 9. PMID 31178433

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin Alone: Metformin was titrated beginning at 500 mg/day to the maximum dose tolerated (up to 2000 mg/day).
- Glargine Followed by Metformin: Basal insulin glargine was titrated to achieve a morning fasting blood glucose of 85-95 mg/dl and continued through 3 months after which metformin was titrated as in the Metformin alone arm and continued for 9 months.
Period: Overall Study
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Started | 47 | 44
Completed | 45 | 41
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Total
Number analyzed (Participants) | 47 | 44 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 42 | 89
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.9 (2.1) | 14.9 (2.0) | 14.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 65
  Male | 9 | 17 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic white | 12 | 13 | 25
  Black | 9 | 14 | 23
  Hispanic | 20 | 14 | 34
  All othe | 6 | 3 | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.9 (6.4) | 36.5 (6.4) | 36.7 (6.4)
HbA1c [Mean (Standard Deviation); unit: % of glycosylated hemoglobin] | 5.7 (0.6) | 5.7 (0.6) | 5.7 (0.6)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 109.2 (19.7) | 107.5 (14.1) | 108.3 (17.1)
2-hour OGTT glucose [Mean (Standard Deviation); unit: mg/dl] | 184.2 (50.2) | 183.5 (44.5) | 183.9 (47.3)

OUTCOME MEASURES:

1. Primary Outcome: ß-cell Response Measured by Hyperglycemic Clamp
Description: Clamp measures of ß-cell response, co-primary outcomes
Time Frame: 3-months after medication washout (Month 15)
Population: Primary analysis was on all participants able to have a M15 visit. 2 participants in the metformin alone arm decompensated at M12 and were unable to remain off treatment until M15. A sensitivity analysis including these 2 participants using 1/2 of the worst value among all other participants did not alter the results.
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Number analyzed (Participants) | 43 | 41
nmol/L
  Steady State C-peptide | 4.82 [2.07 to 11.23] | 4.18 [1.74 to 10.08]
  ACPRmax | 6.92 [2.81 to 17.03] | 5.95 [2.17 to 16.37]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin; Seemingly unrelated regression was used to compare treatment arms on the combination of insulin sensitivity (M/I as calculated from the hyperglycemic clamp) and insulin secretion (steady-state C-peptide and ACPRmax as co-primary; ACPRg as major secondary,). See statistical analysis plan for further details and R code; Test type: Superiority; p > 0.05, Regression, Linear — All analyses were conducted with values on a log scale and re-exponentiated for presentation; Measures of ß-cell response were modeled simultaneously with insulin sensitivity (M/I) using 2-df seemingly unrelated regression models

2. Primary Outcome: M/I
Description: Clamp measure of insulin sensitivity
Time Frame: 3-months after a medication washout
Population: All participants with a Month 15 visit
Measure: Mean (95% Confidence Interval); unit: x 10-5 mmol/kg/min per pmol/L
Groups:
- Metformin Alone: Metformin will be titrated to the maximum dose tolerated (up to 2000 mg/day).
  Metformin
- Glargine Followed by Metformin: Basal insulin glargine for 3 months titrated to achieve a morning fasting blood glucose of 85-95 mg/dl, followed by metformin (titrated up to 2000 mg/day) for 9 months.
  Metformin
  Glargine
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Number analyzed (Participants) | 43 | 41
x 10-5 mmol/kg/min per pmol/L | 1.48 [0.29 to 7.63] | 1.70 [0.25 to 11.54]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin; Analyses were completed on a log scale and re-exponentiated for presentation; Test type: Superiority; p > 0.05, Regression, Linear

3. Secondary Outcome: ACPRg
Description: First phase response
Time Frame: 3-months after a medication washout
Population: Primary analysis was on all participants able to have a M15 visit.
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Number analyzed (Participants) | 43 | 41
nmol/L | 1.11 [0.14 to 8.56] | 1.12 [0.15 to 8.35]

4. Secondary Outcome: ß-cell Function Measured by Hyperglycemic Clamp Techniques at M12
Description: Participants had 12-months of active therapy. Secondary results at the end of active intervention.
Time Frame: End of active intervention (Month 12).
Population: Secondary analysis was on all participants with a Month 12 visit.
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Number analyzed (Participants) | 45 | 41
nmol/L
  Steady State C-peptide | 4.78 [2.09 to 10.94] | 4.37 [1.75 to 10.94]
  ACPRmax | 6.95 [3.16 to 15.28] | 5.79 [2.49 to 13.46]
  ACPRg | 1.06 [0.10 to 11.33] | 1.03 [0.05 to 21.73]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin; Analyses were completed on a log scale and re-exponentiated for display; Test type: Superiority; p > 0.05, Regression, Linear

5. Secondary Outcome: Clamp Measure of Insulin Sensitivity
Description: Participants had 12-months of active therapy. Secondary results at the end of active intervention.
Time Frame: End of active intervention (Month 12)
Population: Secondary analysis was on all participants with a Month 12 visit.
Measure: Mean (95% Confidence Interval); unit: x 10-5 mmol/kg/min per pmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin
Number analyzed (Participants) | 45 | 41
x 10-5 mmol/kg/min per pmol/L | 1.52 [0.17 to 13.48] | 1.93 [0.30 to 12.50]

6. Other Pre Specified Outcome: OGTT Measures of ß-cell Function and Glucose Tolerance
Description: Measures derived the OGTT at the end of the 12 month active intervention period, and following a 3-month and 9-month washout.
Time Frame: After 12 months of active treatment, and 3 and 9 months of washout
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the 21 month study period
Description: AEs were captured at quarterly clinical visits and SAEs were captured as they occur or when reported at a subsequent clinical visit
Arm/Group | Metformin Alone | Glargine Followed by Metformin
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/44
Serious Adverse Events (participants affected / at risk) | 5/47 | 2/44
Other Adverse Events (participants affected / at risk) | 30/47 | 30/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Alone (N=47) | Glargine Followed by Metformin (N=44)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Ewing's Sarcoma
Mental health hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Suicide ideation
Appendicitis (General disorders) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tonsillectomy & Adenoidectomy (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Pnemonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin Alone (N=47) | Glargine Followed by Metformin (N=44)
Low blood sugar (Endocrine disorders) | 0 | 16 — self monitored blood glucose <70 mg/dl during 3 months of glargine treatment
Skin rash (Skin and subcutaneous tissue disorders) | 6 | 6
GI Discomfort (Gastrointestinal disorders) | 16 | 17
Polyuria or polydipsia (Endocrine disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT01779375/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT01779375/SAP_002.pdf
  • Informed Consent Form (2013-05-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT01779375/ICF_001.pdf